CLINICAL TRIAL: NCT07103317
Title: Comprehensive COROnary PHYSiology Assessment in Patients With Angina With Nonobstructive Coronary Arteries - CZECH Republic (CoroPhys-CZECH)
Brief Title: Comprehensive Coronary Physiology in Patients With Angina With Nonobstructive Coronary Arteries - Czech Republic
Acronym: CoroPhys-CZ
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Motol (Other)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other); Nemocnice AGEL Trinec-Podlesi a.s. (Other); Brno University Hospital (Other); Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Petr Kala, MD, Physician, Principal Investigator, University Hospital, Motol
Other Study IDs: EK -151.42/25
Record Dates: First submitted 2025-07-16; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: ANOCA; ANOCA - Angina With Non-obstructive Coronary Arteries; MINOCA; Microvascular Dysfunction; Microvascular Angina; Vasospastic Angina; Acetylcholine
Keywords: ANOCA; INOCA; MINOCA; Coronary Microvascular Dysfunction; Microvascular Angina; Vasospastic Angina; Acetylcholine Testing; Coronary Termodilution
MeSH Terms: conditions — MINOCA; Microvascular Angina; Angina Pectoris, Variant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Biospecimen Retention: Samples Without DNA — Blood - plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronary artery disease (CAD) is a leading cause of morbidity and mortality. While cardiologists have been focused on discrete, visible stenoses of coronary arteries, there is increasing awareness of the importance of microcirculation and vasospastic disorders in causing angina. The microvascular bed is composed of vessels smaller than 400 microns in diameter. Their network is significantly larger than that of the epicardial vessels and serves essential functions, including regulating myocardial blood flow and cellular metabolism.

Angina pectoris, a most frequent symptom of CAD or myocardial ischemia, was assumed to be caused by significant stenosis of the epicardial coronary artery. However, it was found that in over 50% of cases, there was no obstructive CAD, which is described as angina with no obstructive coronary arteries (ANOCA) or ischemia with no obstructive coronary arteries (INOCA), according to the clinical setting.

DETAILED DESCRIPTION:
Two mechanisms are primarily involved in the pathophysiology: structural and functional impairment, which can affect both epicardial and microcirculatory arteries and may also be combined. Thus, from a clinical point of view, two basic endotypes are distinguished in ANOCA: 1) microvascular angina (MVA) due to structural damage of microcirculation (coronary microvascular dysfunction - CMD), or functional microvascular vasospasm (angina and ECG changes without epicardial vasospasm on acetylcholine testing) and 2) epicardial vasospastic angina (VSA) - angina, ECG changes and vasospasm on acetylcholine testing (Table 1).

1. Microvascular Angina (MVA) (FFR > 0,80, iFR > 0,89)

   * coronary microvascular dysfunction (CMD) (CFR < 2,0 (2,5), MRR < 2,1, IMR > 25)
   * microvascular vasospasm (angina + ECG changes + < 90% epicardial spasm during Ach testing)
2. Vasospastic Angina (VSA) (angina + ECG changes + > 90% epicardial spasm during Ach testing)
3. Non-coronary chest pain (negative thermodilution and Ach testing)

Table 1 - ANOCA endotypes. FFR - fractional flow reserve, iFR - instantaneous wave-free ratio, CFR - coronary flow reserve, MRR - microvascular resistance reserve, IMR - index of microcirculatory resistance, EKG - electrocardiogram, Ach - acetylcholine.

The clinical manifestation of ANOCA includes a wide range of symptoms that reduce the quality of life and are often misdiagnosed, mistreated, and not infrequently, leading to repeated hospitalizations and invasive investigations. At the same time, patients with both MVA and VSA have a poorer long-term prognosis. Direct assessment of the response of the coronary microcirculation to vasodilator stimuli and diagnosis of vasomotor abnormalities are crucial for accurate stratification and selection of treatment strategies for patients with ANOCA, resulting in reduced angina severity and improved quality of life compared to standard care. Comprehensive invasive coronary functional testing (CFT) is currently the only diagnostic method to establish a definitive diagnosis and characterize a specific ANOCA endotype, supported by professional societies' current recommendations.

CFT consists of a complete invasive assessment of epicardial and microcirculatory structural and functional disorders. It starts with coronary angiography (CA) to exclude structural epicardial CAD accompanied by testing of the hemodynamic significance of epicardial stenoses by a hyperemic or non-hyperemic index (i.e., fractional flow reserve (FFR) or instantaneous wave-free ratio (iFR)) if necessary. When there is no significant epicardial CAD, the protocol continues with coronary thermodilution to investigate microcirculatory function by measuring intracoronary blood flow and resistances by temperature-pressure intracoronary wire (PressureWire X, Abbott) during rest and hyperemia caused by saline solution infused by a dedicated microcatheter (RayFlow, HexaCath). Coroventis software calculates the coronary flow reserve (CFR) and microvascular resistance reserve (MRR) or index of microcirculatory resistance (IMR) when using bolus thermodilution. CMD occurs when CFR and MRR are reduced, or IMR is increased (Table 2). The last part of the CFT aims to test coronary vasoreactivity to an intracoronary bolus of Acetylcholine (Ach), which should cause vasodilatation in physiological circumstances; however, it may lead to vasoconstriction and vasospasm if endothelial dysfunction or imbalance between vasodilatation and vasoconstriction vascular pathways. The Ach test is positive for VSA when Ach induces symptoms typical for the patient (the reason for the invasive examination), ischemic EKG changes, and proven epicardial spasm by angiography after Ach bolus. When there are only typical symptoms and ischemic EKG changes, but without visible epicardial spasms on angiography, it is concluded as microvascular vasospasm (a sub-endotype of MVA). When all three parts of CFT are negative (CA for epicardial structural CAD, thermodilution for microvascular structural CAD, and Ach testing for vasospasm), the symptoms are suggested to be non-coronary or non-cardiac.

Abbreviation Parameter Methodology Pathology Calculation

1. CFR coronary flow reserve intracoronary Doppler, thermodilution < 2,0-2,5 Doppler: APVhyper/APVrest bolus thermodilution: Tmn,rest/Tmn,hyper cont. thermodilution: Qhyper/Qrest
2. IMR index of microcirculatory resistance bolus thermodilution > 25 Pd x Tmn during hyperemia
3. MRR microvascular resistance reserve continuous thermodilution < 2,1 (CFR/FFR) x (Pa,rest/ Pa,hyper) (Qhyper/Qrest) x (Pa,rest / Pd,hyper)
4. Rmikro absolute resistance continuous thermodilution > 500 WU Pd/Q

Table 2 - Microcirculatory indexes. CFR - coronary flow reserve, MRR - microvascular resistance reserve, IMR - index of microcirculatory resistance, Rmikro - absolute resistance, APV - average peak velocity, Tmn - mean transit time, Q - flow, Pd - distal pressure, FFR - fractional flow reserve, Pa - aortic pressure, WU - Wood Units.

Given all the evidence outlined above, a hypothesis has been formulated:

Specific ANOCA endotypes differ in prevalence, clinical presentation, and therapeutic management. A tailored approach based on leading pathophysiology would improve symptoms and quality of life. EAT plays an important role in the development and pathophysiology of CMD and vasospastic disorders.

The aim is to evaluate the practice of patient selection for the assessment of ANOCA endotypes, including indications, ischemia tests performed, medications prescribed, procedural aspects of microcirculation, and changes in evaluation and treatment following testing. Additionally, investigators seek insight into adverse cardiovascular events in these patients following invasive coronary physiology. Furthermore, the aim is to investigate the pathophysiology of microvascular dysfunction and coronary vasospastic disorders, specifically the relationship between EAT measured by CMR and CMD measured by invasive hemodynamic techniques.

Within this aim, the following specific goals will be addressed:

Aim 1: To assess the practice of patient selection for assessment of invasive coronary physiology, including vasospasm testing and estimation of microcirculation by measuring CFR and IMR or MRR.

Aim 2: To assess procedural aspects of invasive coronary physiology - how parameters mentioned above are measured in the catheterization laboratory.

Aim 3: To assess patients' treatment and changes after invasive coronary physiology measurements at each follow-up visit.

Aim 4: To compare the cardiovascular outcomes and additional procedures (stress testing, angiography, etc.) done after comprehensive invasive coronary physiology evaluation.

Aim 5: To correlate the volume of EAT measured by CMR with results of CFT, especially CFR, MRR, IMR, and vasospasms.

To address these specific goals, the investigators plan to employ the following experimental models and the following drugs.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes older than 18 years
* Angina symptoms or angina equivalent
* Referred to cath lab for evaluation of CAD
* Invasive physiology testing performed (microcirculation testing +/- vasospasm testing)

Exclusion Criteria:

* Persons under the age of 18
* Pregnant of nursing
* No coronary physiology measurements were performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The prospective and observational study will include patients who underwent microcirculation assessment or vasospastic testing using intracoronary Ach (or both as parts of CFT). As described above, participants will undergo routine coronary angiography and comprehensive physiologic testing by coronary thermodilution to evaluate CMD and provocative Ach testing for diagnosing vasospastic angina (VSA).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 1 year
  All-cause death
Components of MACE | 1 year
  Cardiovascular death, MI, coronary revascularisation, stroke, hospitalization for heart failure, hospitalization for acute coronary syndrome, repeated coronary angiography

OTHER OUTCOMES:
Angina severity | 1 year
  Seattle Angina Questionnaire - SAQ - 0 to 100 - the higher the less symptoms
  - change in SAQ score from baseline
Quality of life (EQ-5D-5L) | 1 year
  EQ-5D-5L questionnaire; -0.59 to 1, where 1 is the best possible health state
  - change in EQ-5D-5L score from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Petr Kala, M.D., Ph.D., Principal Investigator — University Hospital Motol, Charles University
Locations (1):
- University Hospital Motol, Prague, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: No